CLINICAL TRIAL: NCT03018756
Title: Use of Nebulized Fentanyl in Patients With Mild-to-Moderate Interstitial Lung Disease and Chronic Dyspnea
Brief Title: Nebulized Fentanyl in Patients With Mild to Moderate Interstitial Lung Disease and Chronic Dyspnea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Denis O'Donnell (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DMED-1921-16
Record Dates: First submitted 2016-12-20; First posted 2017-01-12 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Fentanyl; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl Citrate (Active Comparator): Single dose, nebulized 100 mcg fentanyl citrate. This is a double-blind, placebo-controlled, two-period crossover study comparing the effects of a single dose of nebulized 100 mcg fentanyl citrate to that of a placebo (0.9% saline). Treatments will be in randomized order: patients in one study arm will receive fentanyl at the first treatment visit and placebo at the second treatment visit, patients in the other arm will receive placebo first and fentanyl second.
  Interventions: Drug: Fentanyl Citrate
- Placebo (Placebo Comparator): Single dose, nebulized 0.9% saline solution. This is a double-blind, placebo-controlled, two-period crossover study comparing the effects of a single dose of nebulized 100 mcg fentanyl citrate to that of a placebo (0.9% saline). Treatments will be in randomized order: patients in one study arm will receive fentanyl at the first treatment visit and placebo at the second treatment visit, patients in the other arm will receive placebo first and fentanyl second.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl Citrate — 100 mcg fentanyl citrate will be inhaled via nebulizer.
  Other Names: inhaled fentanyl
  Arms: Fentanyl Citrate
Drug: Placebo — 0.9% saline solution will be inhaled via nebulizer
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
Patients with interstitial lung disease (ILD) experience distressing activity-related respiratory discomfort which is challenging to manage therapeutically. Interventions such as pulmonary rehabilitation, collaborative self-management, supplemental oxygen therapy and oral opiate medications, are variably effective and therapeutic responses to each in individual patients are difficult to predict. The purpose of this study is to evaluate the acute effects of inhaled opiate therapy (fentanyl citrate) on breathing discomfort (dyspnea) in individuals with mild-to-moderate ILD, as well as examine the potential mechanisms of dyspnea relief.

DETAILED DESCRIPTION:
Treatment with opioids can improve activity related dyspnea by reducing central respiratory neural drive. Inhaled fentanyl citrate is an opioid that is generally well tolerated and has been shown to effectively relieve respiratory discomfort without causing systemic side-effects, although its mechanism of action are poorly understood. Based on the current evidence, non-sedating, rapidly active inhaled fentanyl represents a possible alternative and effective treatment of severe dyspnea in patients with ILD who require urgent treatment. As such, the primary objective of this study is to examine the acute effects of nebulized fentanyl on dyspnea intensity and quality in patients with mild-to-moderate ILD, as well as examine the neurophysiological mechanisms of dyspnea relief during fentanyl inhalation. It is believed that fentanyl when compared with placebo, will reduce inspiratory neural drive to the diaphragm and breathing frequency, resulting in improvements in dyspnea intensity during physical exertion. Alternatively, dyspnea relief after inhaled fentanyl may be independent of changes in neural drive, and instead linked to the presence of opioid receptors in the lungs that modulate afferent inputs to the brain, thereby favourably influencing perceived dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Fibrotic interstitial lung disease (ILD) diagnosis confirmed by specialty ILD clinic
* A total lung capacity (TLC) <lower limit of normal and ≥60%predicted, a forced vital capacity (FVC) <lower limit of normal and ≥60%predicted, and a forced expiratory volume in 1 second (FEV1)/FVC >70%.
* Clinically stable as defined by no changes in medication dosage or frequency of administration with no exacerbations or hospital admissions in the preceding 6 weeks.
* Moderate-to-severe chronic activity related dyspnea as defined by a Baseline Dyspnea Index total score ≤9, modified Medical Research Council score >1, or oxygen cost diagram.
* Ability to perform all study procedures and provide/sign informed consent.

Exclusion Criteria:

* Women of childbearing age who are pregnant or trying to become pregnant.
* Diffusing capacity of the lung for carbon monoxide (DLCO) <40 %predicted.
* Presence of active cardiopulmonary disease other than ILD that could contribute to dyspnea and exercise limitation.
* History of allergy or adverse reaction to fentanyl.
* History of allergy or adverse reaction to latex
* Presence of contraindications to pulmonary function or clinical exercise testing, including inability to exercise because of neuromuscular or musculoskeletal disease(s).
* Use of ambulatory oxygen or exercise-induced oxygen desaturation to < 80% on room air.
* Body mass index (BMI) <18.5 or ≥35.0 kg/m2.
* Use of antidepressant drugs (i.e., monoamine oxidase inhibitors, serotonin reuptake inhibitors) in the previous 2 weeks.
* Use of opioid drugs (e.g., morphine, fentanyl, oxycodone, codeine, etc.) in the previous 4 weeks.

Note: Healthy volunteers will only be used to assist in the characterization of the IPF study group, i.e., for comparison of baseline exercise responses. They will not undergo treatment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Dyspnea intensity measured by the 10-point Borg Scale at a standardized time during cycle ergometer exercise | 10-minutes post-treatment
  The 10-point Borg scale ranges from 0 "nothing at all" to 10 "maximal/extremely strong" and will be used to rate the intensity of dyspnea during exercise: a decrease in this rating signifies an improvement. Dyspnea intensity will be assessed at a standardized time (4-minutes) in both post-treatment constant-load cycle ergometer tests.

SECONDARY OUTCOMES:
Diaphragm electromyography (EMGdi) at a standardized time during cycle exercise | 10-minutes post-treatment
  EMGdi will be used as an index of inspiratory neural drive. Assessments will be compared at a standardized time (4-minutes) during both post-treatment constant-load cycle exercise tests.
Ventilation at a standardized time during cycle exercise | 10-minutes post-treatment
  Exercise measurements of minute ventilation will be compared at a standardized time (4-minutes) during both post-treatment constant-load cycle exercise tests.
Breathing frequency at a standardized time during cycle exercise | 10-minutes post-treatment
  Exercise measurements of breathing frequency (respiratory rate) will be compared at a standardized time (4-minutes) during both post-treatment constant-load cycle exercise tests.
Tidal volume at a standardized time during cycle exercise | 10-minutes post-treatment
  Exercise measurements of tidal volume will be compared at a standardized time (4-minutes) during both post-treatment constant-load cycle exercise tests.
Inspiratory capacity at a standardized time during cycle exercise | 10-minutes post-treatment
  Exercise measurements of inspiratory capacity will be compared at a standardized time (4-minutes) during both post-treatment constant-load cycle exercise tests.

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University
Locations (1):
- Respiratory Investigation Unit, Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No